CLINICAL TRIAL: NCT03734731
Title: Clinical Trial Policy Study for the Objective Comparison of Cannabis Vs Opioids (CVO) Pain Management and Therapy Types for Circulatory and Chronic Pain Issues
Brief Title: Cannabis Vs Opioids Pain Management Objective Testing Comparisons
Acronym: CVO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American Association of Sensory Electrodiagnostic Medicine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTSC110118
Record Dates: First submitted 2018-10-23; First posted 2018-11-08 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain; Circulatory Disorders
MeSH Terms: conditions — Chronic Pain | interventions — Transcutaneous Electric Nerve Stimulation; Analgesics, Opioid; nabiximols

STUDY DESIGN:
Intervention Model Description: Individual physician patient studies with all products and services being used on FDA label. Study process being referred to in NCD 310.1 as Clinical Trial Policy (CTP), will be approved by the Principal Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Objective Nerve Conduction testing (Other): Therapy of chronic pain and swelling with Monochromatic Infrared Photo Energy (MIRE) in combination with Transcutaneous Electrical Nerve Stimulation (TENS) and Cannabis or Opioids, to determine which treatment is deemed as the most successful, through objective nerve conduction testing with Neural Scan or AXON-II testing systems. Other types of therapies may be introduced during comparison reviews.
  Interventions: Device: Monochromatic Infrared Photo Energy (MIRE); Device: Transcutaneous Electrical Nerve Stimulation; Drug: Opioids; Drug: Cannabis

INTERVENTIONS:
Device: Monochromatic Infrared Photo Energy (MIRE) — Apply Monochromatic Infrared Photo Energy (MIRE) to the affected nerve
Device: Transcutaneous Electrical Nerve Stimulation — Apply Transcutaneous Electrical Nerve Stimulation (TENS) to the affected nerve
Drug: Opioids — Prescribe Opioids to treat for pain or circulatory disorders, dosage to be determined by Principal Investigator
Drug: Cannabis — Prescribe Cannabis to treat for pain or circulatory disorders, dosage to be determined by Principal Investigator. Comparing Opioid results to Cannabis results with objective nerve testing
  Other Names: Marijuana

SUMMARY:
Our purpose for the study is to find safer, less intrusive, better preforming non-addictive products, as an alternative therapy for pain relief and to help alleviate the opioid epidemic ongoing in America today.

DETAILED DESCRIPTION:
The AASEM nationally Sponsored/ Physicians Clinical Trial Policy CTP (Medicare study) testing results will be concluded by the Principal Investigators (MDs and DOs) of the study at each site authorized to participate by the AASEM, within the highest of scientific mathematical standards, using Pain DX Neural Scan and/or AXON II testing systems, which include amplitude testing certified with Promethius potentiometers, for Small Pain Fiber (SpF) Nerve Conduction Testing, CMS Carrier CPT codes 95904 now 95909 through 95913 units, as needed.

It is expected that, at a later date, other products used for therapy and/or rehabilitation purposes will be added to the comparison protocol for the National Trial Number (NCT# TBA) assigned by the National Library of Medicine (NLM). Other products and/or DME equipment may include: infrared light therapy CPT code 97026, TENS therapy and home units CPT therapy code # 97032, as well as montmorillonite minerals for physical applications (montmorillonite is a natural mineral and has no CPT code - is not a CMS ordinarily payable event).

ELIGIBILITY:
Inclusion Criteria:

* In the investigator's judgment a high probability of 5 year survival.
* Patient is able to comply with the study visit schedule.
* Patient has the ability to comprehend and sign an informed consent document prior to study enrollment.

Exclusion Criteria:

* In the investigator's judgment not a high probability of 5 year survival.
* Patient is unable to comply with the study visit schedule.
* Patient does not have the ability to comprehend and sign an informed consent document prior to study enrollment.

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-06-03 (Estimated); Primary Completion 2027-02-03 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in pain and swelling, as verified by objective nerve conduction testing | 4 to 8 weeks per nerve
  To note changes in axon nerve firings obtained by nerve amplitude measurements. Categorize pain and swelling disorders' treatment success or failure, as defined within the AASEM, using the Neural Scan or AXON-II objective nerve conduction testing systems, with objective responses

CONTACTS AND LOCATIONS:
Overall Officials: Ronald F Davis, Study Director — AASEM/ADAPT/DTSC; Brook Davis, Study Director — ADAPT/DTSC; James Hedgecock, D.C., PhD, Study Director — American Association of Sensory Electrodiagnostic Medicine; Chad Pfefer, M.D., Study Chair — American Association of Sensory Electrodiagnostic Medicine; Michael F Boyer, M.D., Principal Investigator — American Association of Sensory Electrodiagnostic Medicine

IPD SHARING:
Plan to Share IPD: Yes
Through AASEM publications
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Annually reviews / new CME training course provided periodically during every year
Access Criteria: Must be an AASEM certified physician/principal investigator or trial personnel. Otherwise may be obtained on AASEM website.